CLINICAL TRIAL: NCT05226273
Title: Occupational Exposure to Dust and the Relationship With the Respiratory Symptoms, Lung Function Among Construction Workers of the University of Malaysia Sabah (UMS)
Status: Completed | Type: Observational
Sponsor: Universiti Malaysia Sabah (Other)
Responsible Party: Principal Investigator, Abdul Rahman Ramdzan, Clinical Dr, Principal Investigator, Universiti Malaysia Sabah
Other Study IDs: JKEtika 3/18 (9).
Record Dates: First submitted 2022-01-25; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Occupational Exposure
Keywords: Occupational exposure, Air pollution, Lung function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Background The respiratory tract often becomes the site of injury from occupational exposure. All construction sites generate high levels of dust, typically from concrete, silica, asbestos, cement, wood, stone, sand and therefore, the workers are exposed to this airborne dust and increased their risk of developing respiratory disorders. Limited studies have been conducted to assess the relationship between respiratory symptoms, lung function and occupational dust exposure among construction workers in Sabah. The objectives of this study are to determine the occupational exposure to dust and the relationship with the respiratory symptoms as well as lung function among construction workers in UMS Teaching Hospital.

Materials and methods This cross-sectional study consisted of construction workers working in all sections in the development of UMS Teaching Hospital. A standard respiratory questionnaire was distributed to construction workers and lung function measurement was performed using Spirometry and the results of their respiratory status were compared between workers who were exposed and unexposed to dust. Occupational dust exposure was determined by the gravimetric method using an air sampler. The total duration of the collection was 8 hours and the filters with the dust samples were analyzed in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* all construction worker

Exclusion Criteria:

* has chronic lung impairment

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: construction workers who work at the construction site
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Occupational exposure to dust | 2019-2020
  Number of participants with Occupational exposure to dust and having respiratory symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaysia Sabah, Kota Kinabalu, Sabah, Malaysia